CLINICAL TRIAL: NCT04974008
Title: An Open-Label Phase 2 Study of Maintenance Therapy With OST31-164 After Resection of Recurrent Osteosarcoma
Brief Title: Osteosarcoma Maintenance Therapy With OST31-164
Acronym: OST-164-01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emerald Clinical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OST31-164-01 (AOST2121)
Record Dates: First submitted 2021-07-01; First posted 2021-07-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Bone Cancer
Keywords: Osteosarcoma; Bone Cancer
MeSH Terms: conditions — Bone Neoplasms; Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OST31-164 (Experimental): Patients who will receive OST31-164 as a single agent every 3 weeks for 48 weeks with 4 doses constituting 1 treatment cycle (12 weeks per cycle). Each patient will receive treatment at a dose of 1x109 CFU until week 48 or until disease progression, unacceptable toxicity, or the patient meets any other treatment discontinuation criteria.
  Interventions: Drug: OST31-164

INTERVENTIONS:
Drug: OST31-164 — Patients who will receive OST31-164 as a single agent every 3 weeks for 48 weeks with 4 doses constituting 1 treatment cycle (12 weeks per cycle). Each patient will receive treatment at a dose of 1x109 CFU until week 48 or until disease progression, unacceptable toxicity, or the patient meets any other treatment discontinuation criteria.

SUMMARY:
Up to 45 Patients aged 12 to 39 with osteosarcoma (bone cancer) that had recurred in the lungs and has recently been surgically removed will be enrolled. Patients will receive OST31-164 infusions every 3 weeks over 48 weeks and be followed after that for 3 years.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, multicenter, single-arm study in patients (12-39 years) with a recent history of pulmonary recurrent osteosarcoma that has been completely resected. Planned enrollment is a maximum of 45 patients who will receive OST31-164 as a single agent every 3 weeks for 48 weeks with 4 doses constituting 1 treatment cycle (12 weeks per cycle). Each patient will receive treatment at a dose of 1x109 CFU until week 48 or until disease progression, unacceptable toxicity, or the patient meets any other treatment discontinuation criteria. Following treatment discontinuation, all patients will enter a 3-year survival follow-up period. Exploratory evaluation of immune response will be conducted. If available, tissue from the recent resection will be sent to the COG Biobank for future genomic and pathologic analysis by the COG.

ELIGIBILITY:
Inclusion Criteria:

* Note: Patients enrolled on AOST2031 are eligible for enrollment in the present study.

Patients are eligible to be included in the study only if all the following criteria apply:

Age and Weight

1. Between 12 years of age and 39 years of age at the time the Informed Consent/ Assent form is signed.
2. Weight at least 40 kg. Diagnosis
3. Has histologic confirmation of osteosarcoma at diagnosis.
4. Has at least one episode of disease recurrence in the lungs without limitation on the number of episodes of recurrence as long as the following criteria are met:

   1. Surgical resection of all possible sites of suspected pulmonary metastases to achieve a complete remission within 8 weeks prior to study enrollment
   2. Pathological confirmation of osteosarcoma from at least one resected tumor.
   3. Patients will not require radiographic confirmation of complete remission for enrollment. However, a postoperative CT chest scan is required as a baseline for future comparisons.

   https://members.childrensoncologygroup.org/files/Disc/surgery/handbooks/OsteoBoneHandbook.pdf) Performance Status
5. Patient must have a performance status corresponding to ECOG scores of 0, 1, or 2. Use Karnofsky scale for patients > 16 years of age and Lansky scale for patients < years of age Prior Therapy
6. Patient must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, radiotherapy, or surgery prior to entering this study.

   Organ Function Requirements
7. Patient has adequate organ function as defined below:

   a. Hematological: i. Absolute neutrophil count (ANC) is at least 1,000/µL without transfusion or growth factor support. ii. Platelet count ≥ 50,000/µL without transfusion or growth factor support. b. Adequate renal function defined as: i. Creatine clearance or radioisotope glomerular filtration rate (GFR) > 70 mL/min/1.73 m2 or ii. A serum creatine based on age/gender as follows:

   Maximum Serum Creatinine (mg/dL)

   Age: 12 to < 13 years Male :1.2 Female:1.2 Age:13 to < 16 years Male :1.5 Female:1.4 Age: ≥ 16 years Male :1.7 Female:1.4 Note: the threshold for creatinine values in this table were derived from the Schwartz formula for estimating GFR.

   c. Adequate liver function defined as: i. Total bilirubin < 1.5 x upper limit of normal (ULN) for age ii. Serum glutamic-pyruvic transaminase (SGPT) / alanine aminotransferase (ALT) < 110 U/L (for the purpose of this study the ULN for SGPT is 45 U/L) iii. Serum albumin > 2 g/dL

   d. Adequate coagulation i. International normalized ratio (INR) or prothrombin time (PT) < 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or INR is within therapeutic range of intended use of anticoagulants.

   ii. Activated partial thromboplastin time (aPTT) < 1.5 x ULN unless patient is receiving anticoagulant therapy as long as aPTT is within therapeutic range of intended use of anticoagulants.

   e. Adequate cardiac function defined as: i. Shortening fraction of > 27% by echocardiogram, or ii. Ejection fraction of > 50% by radionuclide angiogram or echocardiogram f. Adequate pulmonary function defined as: i. No evidence of dyspnea at rest, no history of exercise intolerance, and a pulse oximetry of > 94%.

   g. Central nervous system (CNS) function defined as: i. Patients with a known seizure disorder may be enrolled if on anticonvulsants and/or are well-controlled.

   ii. CNS toxicity including peripheral neuropathy < Grade 2.
8. Patient and/or patient's parent or legal guardian must be capable of understanding the investigational nature, potential risks, and benefits of the study. The patient and/or the parent or legal guardian must sign a written informed consent. Age-appropriate assent will be obtained per institutional guidelines.

   Contraception:

   Female patients :
9. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in the protocol OR
   2. A WOCBP who agrees to follow the contraceptive guidance in the protocol during the treatment period and for at least 120 days after the last dose of study treatment.
10. A female patient of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving any dose of study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

    Male patients:
11. A male patient is eligible to participate if he agrees to follow the contraceptive guidance in the protocol during the study treatment period and for at least 120 days after the last dose of study treatment.

Exclusion Criteria:

1. Has clinically evident metastatic or recurrent disease.
2. Has concurrent pulmonary recurrence and local recurrence at the primary tumor site.
3. Has primary refractory disease with progression of the primary tumor on initial-therapy.
4. Has CNS or any extrapulmonary disease involvement at the time of the most recent episode of disease recurrence proceeding enrollment.
5. Has active infection requiring systemic therapy or is dependent on or is currently receiving systemic antibiotics that cannot be discontinued before dosing. (Note: Patients who discontinue an antibiotic prior to dosing must wait at least 5 half-lives after the last dose of antibiotic before receiving any OST31-164 infusion). Inhaled prophylactic PJP (pneumocystis jiroveci pneumonia) treatment is acceptable per Investigator discretion.
6. Is currently dependent on or has received corticosteroids within the past 4 weeks (topical corticosteroids and occasional inhaled corticosteroids are allowed).
7. Is currently participating in or has participated in a study of an investigational agent or is using an investigational device within 4 weeks of the first dose of treatment.
8. Has a history of other active malignancy for < 2 years prior to enrollment. Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy or is felt by the Investigator to be at low risk for recurrence is allowed.
9. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients who require intermittent use of bronchodilators or local steroid injections will not be excluded from the study. Patients with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment.
12. Has a known allergy to any component of the study treatment(s) formulations.
13. Has a contraindication (e.g., sensitivity/allergy) to both trimethoprim/ sulfamethoxazole and amoxicillin.
14. Has contraindication to administration of NSAIDs.
15. Is currently receiving or will be receiving any chemotherapy, including PI3K inhibitors, during the treatment phase.
16. Has had a prior monoclonal antibody therapy within 2 weeks prior to study Day 1.
17. Requires or anticipates requiring tumor necrosis factor (TNF) blocking agent (e.g., infliximab) therapy for diagnosis of rheumatologic disease or inflammatory bowel disease (e.g., ankylosing spondylitis, Crohn's disease, plaque psoriasis, psoriatic arthritis, rheumatoid arthritis, or ulcerative colitis).
18. Has previous history of listeriosis.
19. Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
20. Has known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected).
21. Has received a live vaccine within 30 days prior to Study Day 1.
22. Patient is or has an immediate family member (spouse, children, or parent) who is directly involved with this study or is employed by the investigational site or Sponsor, unless prospective Institutional Review Board (IRB) approval (by chair or designee) is given allowing exception to this criterion for a specific patient.

Regulatory Requirements:

1. All patients and/or their parents or legal guardians must sign a written informed consent.
2. All institutional, FDA, and NCI requirements for human studies must be met.

Ages: 12 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival | Every 3 months, up to one year
  The relative proportion of patients experiencing event-free (recurrence-free) survival at 12 months, compared to historical controls. Patients will be e valuated for recurrence every 3 months, consistent with the standard of care.

SECONDARY OUTCOMES:
Overall Survival | Every 3 months, up to 3 years
  Overall survival of patients for three years will be compared to the 3-year overall survival of historical controls. Patients will be followed every 3 months for overall survival for 3 years.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Throughout the treatment period of 48 weeks, then every 3 months for 3 years
  Incidence of Treatment-Emergent Adverse Events as assessed by NCI CTCAE 5.0. Safety will be assessed throughout the treatment period of 48 weeks. Assessments of potential persistence of the vector every 3 months, will continue for an additional 3 years after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Petit, PhD, Study Director — OS Therapies, Inc.
Locations (21):
- United States (21):
  - Kaiser Permanente Downey Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Connecticut Children's, Hartford, Connecticut
  - Nemours/ Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No